CLINICAL TRIAL: NCT00003616
Title: Phase I/II Trial of Irinotecan (CPT-11) in Patients With Recurrent Malignant Glioma
Brief Title: Irinotecan in Treating Patients With Progressive or Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTC-9801; CDR0000066694 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult brain stem glioma; adult oligodendroglioma; adult mixed glioma; adult diffuse astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Oligodendroglioma; Glioma; Astrocytoma | interventions — Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I/II trial to study the effectiveness of irinotecan in treating patients who have progressive or recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and the dose limiting toxicities of irinotecan in patients with progressive or recurrent malignant glioma. II. Define the safety profile of every 3 week dosing of irinotecan in these patients. III. Characterize the pharmacokinetic profile of this regimen in these patients. IV. Assess evidence of antitumor activity in these patients. V. Determine the efficacy of irinotecan in these patients as measured by 6 month progression-free survival and objective tumor response. VI. Evaluate further the safety profile of irinotecan in these patients during phase II study.

OUTLINE: This is a dose escalation study. Patients are stratified according to concurrent enzyme-inducing antiepileptic drugs (EIAEDs)(yes vs no). Group A (without EIAEDs): Patients receive irinotecan IV over 90 minutes on day 1, followed by up to 3 weeks of rest. Group B (with EIAEDs): Patients receive the same treatment but dose escalation is performed in cohorts of 3 patients. The maximum tolerated dose (MTD) is defined as the dose below that at which 2 of 6 patients experience dose limiting toxicities. The Phase I MTD is the starting dose recommended for use in the Phase II portion of the study. Treatment continues every 3 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients are followed every 2 months for 1 year, every 3 months for 1 year, every 4 months for 1 year, then every 6 months until disease progression. Patients are then followed every 4 months for survival.

PROJECTED ACCRUAL: Up to 30 patients will be accrued for phase I within 10 months. A total of 48 patients will be accrued for phase II within 6-8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven progressive or recurrent primary malignant glioma Phase I (excluding group A patients): No more than 2 prior chemotherapy regimens, including 1 prior adjuvant therapy and 1 prior regimen for recurrent or progressive tumor, or 2 prior regimens for progressive tumor Phase II and/or group A patients: No more than 1 prior chemotherapy regimen, either as adjuvant or for recurrent disease Measurable disease by MRI or CT scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 3 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No uncontrolled hypertension No unstable angina No symptomatic congestive heart failure No myocardial infarction within 6 months No serious uncontrolled cardiac arrhythmia Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No severe nonmalignant systemic disease or active infection No concurrent alcoholism or drug abuse No psychosis HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy No concurrent sargramostim (GM-CSF) Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, or suramin) No prior irinotecan, topotecan, or other topotecan 1 inhibitors No other concurrent chemotherapy Endocrine therapy: Stable or decreasing dosage of corticosteroids within 72 hours of study entry (phase II only) No other concurrent immunosuppressive agents No concurrent hormonal therapy Radiotherapy: At least 4 weeks since prior radiotherapy Patients with prior interstitial brachytherapy or stereotactic radiosurgery must have confirmation of progressive disease No concurrent radiotherapy Surgery: At least 3 weeks since prior resection Other: Acute toxic effects (excluding neurotoxicity or alopecia) of any prior therapy must be resolved No concurrent valproic acid as a single agent Concurrent enzyme-inducing antiepileptic drugs (EIAED) with or without steroids are allowed No concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-10-22 (Actual); Primary Completion 2002-05-17 (Actual); Study Completion 2005-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prados, MD, Study Chair — UCSF Medical Center at Parnassus
Locations (10):
- United States (10):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Prados MD, Lamborn K, Yung WK, Jaeckle K, Robins HI, Mehta M, Fine HA, Wen PY, Cloughesy T, Chang S, Nicholas MK, Schiff D, Greenberg H, Junck L, Fink K, Hess K, Kuhn J; North American Brain Tumor Consortium. A phase 2 trial of irinotecan (CPT-11) in patients with recurrent malignant glioma: a North American Brain Tumor Consortium study. Neuro Oncol. 2006 Apr;8(2):189-93. doi: 10.1215/15228517-2005-010. Epub 2006 Mar 13. PMID 16533878
- [Result] Prados MD, Yung WK, Jaeckle KA, Robins HI, Mehta MP, Fine HA, Wen PY, Cloughesy TF, Chang SM, Nicholas MK, Schiff D, Greenberg HS, Junck L, Fink KL, Hess KR, Kuhn J; North American Brain Tumor Consortium study. Phase 1 trial of irinotecan (CPT-11) in patients with recurrent malignant glioma: a North American Brain Tumor Consortium study. Neuro Oncol. 2004 Jan;6(1):44-54. doi: 10.1215/S1152851703000292. PMID 14769140